CLINICAL TRIAL: NCT04119895
Title: Does Neuromuscular Electrical Stimulation Have an Additive Effect to Core Stabilization Exercises on Pain, Disability and Ultrasonographic Thickness of Abdominal and Lumbar Muscles in Chronic Low Back Pain?
Brief Title: Neuromuscular Electrical Stimulation in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018.174.IRB1.022
Record Dates: First submitted 2019-04-12; First posted 2019-10-09 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain
Keywords: Electric stimulation; Ultrasonography; Exercise Therapy; Rehabilitation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES and exercise (Experimental): Neuromuscular electrical stimulation and core stabilization exercise
  Interventions: Other: Neuromuscular electrical stimulation and core stabilization exercise
- Sham NMES and exercise (Sham Comparator): Sham neuromuscular electrical stimulation and core stabilization exercise
  Interventions: Other: Sham neuromuscular electrical stimulation and core stabilization exercise

INTERVENTIONS:
Other: Neuromuscular electrical stimulation and core stabilization exercise — In NMES group, the amplitude of the electrical current will be set at the highest level subject can tolerate.
  The lumbar stabilization mode of the device will be used. This mode consists of three phases; warming, contraction and recovery phases. The duration will be set to 35 minutes. In the first 2 minutes (warming phase), frequency is 6 Hz. Contraction phase includes consecutive cycles of contractile frequency of 40 Hz for 6 seconds and the rest frequency of 4 Hz for 12 seconds, lasting a total of 30 minutes. The last 3 minutes (recovery phase) frequency is 3 Hz. The ramp up time is 2 seconds and the ramp down time is 1 second
  Arms: NMES and exercise
Other: Sham neuromuscular electrical stimulation and core stabilization exercise — In sham NMES group, the amplitude of the electrical current will be set at a minimum level which does not stimulate any contraction.
  Arms: Sham NMES and exercise

SUMMARY:
This study evaluates whether there is additive effect of neuromuscular electrical stimulation applied to lower lumbar region to core stabilization exercises in the management of chronic low back pain. Participants will randomly divide into two groups; half will receive core stabilization exercises and neuromuscular electrical stimulation (NMES) in combination, while the other half will receive core stabilization exercises and sham NMES.

DETAILED DESCRIPTION:
Patients with low back pain cannot activate enough the deep lumbar stabilization muscles necessary for spinal stability, such as transversus abdominis, lumbar multifidus.

Core stabilization exercises are valuable in motor relearning of coactivation of deep lumbar and abdominal muscles and in stabilization of the spine. Hence, they are important in the management of chronic low back pain.

Neuromuscular electrical stimulation (NMES) has been used in the training and strengthening of skeletal muscles for many years. It is shown that NMES can contract deep lumbar stabilization muscles and changes in muscle activation are significantly associated with pain reduction in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Pain intensity greater than 3 over 10,
* Pain duration more than 3 months,
* Consent to participate in the study

Exclusion Criteria:

* Previous lumbar surgery,
* Radiculopathy,
* Non-mechanical back pain,
* Acute low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index | 4 weeks (change from baseline to 4 weeks after)
  Oswestry Disability Index (ODI), measures the level of disability. It consists of 10 items questioning the severity of pain, self-care, lifting and carrying, walking, sitting, standing, sleep, the degree of pain change, travel and social life. Its Turkish version is validated in 2004. Items are scored between 0 and 5, and the total score is multiplied by two. The maximum score is "100". As the total score increases, the level of disability increases.

SECONDARY OUTCOMES:
Change in Visual Analog Scale | 4 weeks (change from baseline to 4 weeks after)
  It is a scale consisting of a 10-centimeter line that evaluates the intensity of pain. Starting point of scale, 0 = no pain, end point 10 = expressed as the most severe pain encountered in life. Patients are asked to mark the severity of pain on the line. When calculating, the distance between the marked point and the starting point is measured in centimeters. Increasing the score means that the pain intensity increases.
Change in Nottingham Health Profile | 4 weeks (change from baseline to 4 weeks after)
  Nottingham health profile is a general quality-of-life questionnaire that measures health problems that a person perceives and how these problems affect normal and daily activities. The questionnaire consists of 38 items and evaluates 6 dimensions related to health: energy, pain, emotional reactions, sleep, social isolation and physical activity. Questions are answered as yes or no. Scoring is done in every section between 0-100. 0 indicates the best health status, 100 worst health status. The total Nottingham Health Profile score is obtained from the sum of the sub-scores. Turkish validity and reliability were shown in 2000.
Change in Ultrasonographic thickness of multifidus and abdominal muscles | 4 weeks (change from baseline to 4 weeks after)
  Participants will be asked to lie in supine position with feet flat, knees flexed 90 degree and hips flexed about 45 degrees. Probe is placed transversely at the intersection point of two lines, one horizontal line passing through umbilicus and second vertical line passing through anterior superior iliac spine to visualize the transversus abdominis, oblique internus and oblique externus. No pressure applied. The image is taken at the end of expiration.
  Participants will be asked to lie in prone position with a pillow placed under the abdomen to minimize the lumbar lordosis. Probe will be placed longitudinally over L3, L4, L5 spinous processes with reference to the sacrum and moved to both sides to view the multifidus muscles at these levels in a single screen to measure muscle thickness. Then probe will be placed transversely and moved laterally until the facet joints are seen in the screen to visualize the multifidus muscles and to measure its area at each level.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was not planned to share individual participant data.

REFERENCES:
- [Result] Hoy D, March L, Brooks P, Woolf A, Blyth F, Vos T, Buchbinder R. Measuring the global burden of low back pain. Best Pract Res Clin Rheumatol. 2010 Apr;24(2):155-65. doi: 10.1016/j.berh.2009.11.002. PMID 20227638
- [Result] Kim SY, Kim JH, Jung GS, Baek SO, Jones R, Ahn SH. The effects of transcutaneous neuromuscular electrical stimulation on the activation of deep lumbar stabilizing muscles of patients with lumbar degenerative kyphosis. J Phys Ther Sci. 2016 Jan;28(2):399-406. doi: 10.1589/jpts.28.399. Epub 2016 Feb 29. PMID 27064323
- [Result] Coghlan S, Crowe L, McCarthyPersson U, Minogue C, Caulfield B. Electrical muscle stimulation for deep stabilizing muscles in abdominal wall. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:2756-9. doi: 10.1109/IEMBS.2008.4649773. PMID 19163276
- [Result] Coghlan S, Crowe L, McCarthypersson U, Minogue C, Caulfield B. Neuromuscular electrical stimulation training results in enhanced activation of spinal stabilizing muscles during spinal loading and improvements in pain ratings. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:7622-5. doi: 10.1109/IEMBS.2011.6091878. PMID 22256103
- [Result] Fairbank JC. Oswestry disability index. J Neurosurg Spine. 2014 Feb;20(2):239-41. doi: 10.3171/2013.7.SPINE13288. Epub 2013 Nov 22. No abstract available. PMID 24266676
- [Result] Ohnhaus EE, Adler R. Methodological problems in the measurement of pain: a comparison between the verbal rating scale and the visual analogue scale. Pain. 1975 Dec;1(4):379-384. doi: 10.1016/0304-3959(75)90075-5. PMID 800639
- [Result] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Result] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Result] Hunt SM, McKenna SP, McEwen J, Williams J, Papp E. The Nottingham Health Profile: subjective health status and medical consultations. Soc Sci Med A. 1981 May;15(3 Pt 1):221-9. doi: 10.1016/0271-7123(81)90005-5. No abstract available. PMID 6973203
- [Result] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Result] Liddle SD, Baxter GD, Gracey JH. Exercise and chronic low back pain: what works? Pain. 2004 Jan;107(1-2):176-90. doi: 10.1016/j.pain.2003.10.017. PMID 14715404
- [Result] Akhtar MW, Karimi H, Gilani SA. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial. Pak J Med Sci. 2017 Jul-Aug;33(4):1002-1006. doi: 10.12669/pjms.334.12664. PMID 29067082